CLINICAL TRIAL: NCT05140083
Title: 68Ga-NOTA Evans Blue PET/CT in Patients With Lymphatic System Related Diseases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian13
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Positron-Emission Tomography
Keywords: Lymphatic System Related Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA Evans Blue PET/CT in Patients with Lymphatic System Related Diseases (Experimental): A single dose of 37-111 Mega-Becquerel (MBq) 68Ga-NOTA Evans Blue will be injected subcutaneously. PET/CT imaging will be performed at 5-30 min post- injection. Visual and quantitative method will be used to assess the PET/CT images.
  Interventions: Drug: 68Ga-NOTA Evans Blue

INTERVENTIONS:
Drug: 68Ga-NOTA Evans Blue — Each subject receives a single subcutaneous injection of 68Ga-NOTA Evans Blue, and undergo PET/CT imaging within the specific time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-NOTA Evans Blue (68Ga-NEB) positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and efficacy assessment in lymphatic system related diseases.

DETAILED DESCRIPTION:
Subjects with lymphatic system related diseases underwent 68Ga-NEB PET/CT either for a primary diagnosis or for efficacy assessment. Anomalies were detected by visual analysis and quantitative analysis of maximum standard uptake value (SUVmax). To compare the diagnostic sensitivity of 68Ga-NEB PET/CT lymphatic imaging with other lymphatic imaging such as 99mTc-dextran for lymphatic system related diseases.

ELIGIBILITY:
Inclusion Criteria:

* adult population (aged between18 years and 80 years)
* patients with suspected or new diagnosed or previously treated lymphatic system related diseases
* patients who had scheduled 68Ga-NEB PET/CT scan
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee

Exclusion Criteria:

* patients with pregnancy
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analysis of lymphatic patency | through study completion, an average of 3 years
  The bilateral lymphatic description on 68Ga-NEB PET/CT and lymphatic SPECT imaging were compared. The patency of lymphatic vessels (including lymphatic disruption, dermal distribution, and so on, results are indicated by 0 and 1) are shown in two imagings were recorded respectively.
Standardized uptake value (SUV) | through study completion, an average of 3 years
  Standardized uptake value (SUV) of 68Ga-NEB for each target lesion of subject.

SECONDARY OUTCOMES:
Diagnostic efficacy | through study completion, an average of 3 years
  The sensitivity of 68Ga-NEB PET/CT and lymphatic SPECT imaging were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No